CLINICAL TRIAL: NCT03973125
Title: Application of Intravitreal Conbercept Injection as a Primary Treatment for Exudative Circumscribed Choroidal Haemangioma: Short-term Follow-up of Anatomical and Functional Responses
Brief Title: Application of Intravitreal Conbercept Injection as a Primary Treatment for Exudative Circumscribed Choroidal Haemangioma
Acronym: IVCCCH
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018KYPJ082
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Circumscribed Choroidal Haemangioma
Keywords: circumscribed choroidal haemangioma; conbercept; effectiveness; safety
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The patients in the treatment group receive three monthly intravitreal injection of conbercept followed by PRN rescue treatments such as intravitreal injection of conbercept, laser photocoagulation (when outside the macular) or photodynamic therapy (when in the macular).
  Interventions: Drug: conbercept

INTERVENTIONS:
Drug: conbercept — After three monthly injections of conbercept, if no effects was seen in the patients, the patients will receive rescue treatments such as photodynamic therapy (in the macular) or laser photocoagulation (outside the macular).

SUMMARY:
The aim of this study was to investigate the safety and effectiveness of application of intravitreal conbercept injection as the primary treatment for exudative circumscribed choroidal haemangioma.

DETAILED DESCRIPTION:
This prospective clinical trial aims to evaluate the safety and effectiveness study of intravitreal conbercept injection as the primary treatment for exudative circumscribed choroidal haemangioma: (1)To evaluate therapeutic effect (including both anatomical and functional responses to intravitreal conbercept injection) of intravitreal conbercept injectionfor exudative circumscribed choroidal haemangioma; (2)To evaluate the safety (including side effects of the eye as well as side effects of system) of intravitreal conbercept injection for exudative circumscribed choroidal haemangioma.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients with circumscribed choroidal haemangioma who was diagnosed using ophthalmoscopy, fluorescein/indocyanine green angiography, and ultrasonography; 2) presence of reduced visual acuity or metamorphopsia; and 3) subretinal fluid involving the fovea.

Exclusion Criteria:

* patients with abnormal liver function test results, liver disease, porphyria, or previous treatment for circumscribed choroidal haemangioma.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08-28 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | half a year
  change of best corrected visual acuity

SECONDARY OUTCOMES:
Central foveal thickness | half a year
  change of central foveal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Kunbei Lai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided